CLINICAL TRIAL: NCT04863287
Title: A Phase 1 Study in Healthy Subjects to Evaluate the Safety and Pharmacokinetics of a Human Monoclonal Antibody (2217LS) Against Borrelia Burgdorferi (B. Burgdorferi) Outer Surface Protein A (OspA)
Brief Title: First Clinical Study of the Safety and Blood Levels of a Human Monoclonal Antibody (2217LS) Against Lyme Disease Bacteria in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MassBiologics (Other)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: MBL-LYME-20-01
Record Dates: First submitted 2021-04-14; First posted 2021-04-28 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Lyme Disease
Keywords: LYME; Lyme bacteria; Borrelia burgdorferi (B. burgdorferi); Human Monoclonal Antibody; Outer surface protein A (OspA)
MeSH Terms: conditions — Lyme Disease | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, partial-blind, placebo controlled, sequential, dose escalation study, consisting of four cohorts of 10 subjects. Each cohort will have a sentinel group consisting of 2 subjects randomized 1:1 to receive 2217LS or placebo. Sentinel subjects will be dosed first. If judged safe and well tolerated by the Principal Investigator (PI) and if the stopping rules have not been met, the remaining 8 subjects in the cohort will be randomized 7:1 to 2217LS or placebo, respectively and dosed no less than 24 hours after dosing of sentinel subjects has been completed.
  For each cohort, safety and pharmacokinetic (PK) data will be reviewed by the PI, Independent Medical Monitor (IMM) and Sponsor prior to dosing the next cohort. A minimum of 7 days of safety data and available PK data from a minimum of 8 subjects from the preceding cohort must be reviewed. Dosing of the next cohort may proceed upon agreement between the PI, IMM and Sponsor, if the stopping rules have not been met.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 0.5 mg/kg of 2217LS (Experimental): Single dose subcutaneous injection
  Interventions: Biological: 2217LS
- 1.5 mg/kg of 2217LS (Experimental): Single dose subcutaneous injection
  Interventions: Biological: 2217LS
- 5 mg/kg of 2217LS (Experimental): Single dose subcutaneous injection
  Interventions: Biological: 2217LS
- 10 mg/kg of 2217LS (Experimental): Single dose subcutaneous injection
  Interventions: Biological: 2217LS
- 0.9% Sodium Chloride (NaCl) (Placebo Comparator): Single dose subcutaneous injection
  Interventions: Other: 0.9% Sodium Chloride (NaCl)

INTERVENTIONS:
Biological: 2217LS — Fully Human Monoclonal Antibody
  Arms: 0.5 mg/kg of 2217LS; 1.5 mg/kg of 2217LS; 10 mg/kg of 2217LS; 5 mg/kg of 2217LS
Other: 0.9% Sodium Chloride (NaCl) — Subcutaneous injection
  Arms: 0.9% Sodium Chloride (NaCl)

SUMMARY:
This is a research study of the investigational drug 2217LS in healthy volunteers. Investigational means 2217LS is a new drug that has not been approved for the treatment of any disease. 2217LS is human antibody designed to provide protection from Lyme disease. Lyme disease is a disease carried by infected ticks and can cause the infection to spread to the joints, heart and nervous system in humans.

This is the first time 2217LS will be given to humans. This is not a study of how well 2217LS works against Lyme disease. The only purposes of this study are to: 1) Learn about the safety and tolerability of a subcutaneous (SC [under the skin]) injection of 2217LS when administered to healthy volunteers. 2) Find out how much 2217LS is in the blood of healthy volunteers after receiving 2217LS SC.

In this study, groups of healthy volunteers will be given different doses of 2217LS by SC injection. Volunteers will stay in the study unit for a total of 4 overnights. The planned duration of participation is up to 14 months. Study personnel will monitor their safety using standard procedures like physical examinations, electrocardiograms, questions about possible side effects, blood and urine tests. The amount of 2217LS in their blood will also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent and able to effectively communicate with the Investigator and study personnel. A signed informed consent form (ICF) must be on file prior to initiating the screening procedures.
2. Willing and able to complete all study requirements, restrictions, visits and procedures.
3. Negative for serum anti-B. burgdorferi antibodies by an FDA approved modified two-tier ELISA test.
4. Age 19 to 65 years, inclusive.
5. Weight 50 kg to 105 kg, inclusive.
6. Seated blood pressure is greater than 90/40 mmHg or less than 140/90 mmHg at the screening visit, and seated heart rate is higher than 40 bpm or lower than 99 bpm at the screening visit.
7. Women of reproductive potential must agree not to become pregnant for at least 12 months after the study product administration. If a woman is sexually active and has no history of hysterectomy or tubal ligation, she must agree to use hormonal or barrier birth control with spermicidal gel.
8. Males of reproductive potential must use a barrier method of contraception during the course of the study.
9. Screening laboratory values must meet the following criteria:

   * WBC > 3,900 and < 11,000/mm3
   * Platelets > 100,000/mm3
   * Hemoglobin > 10.5 gm/dl
   * Creatinine ≤ ULN
   * BUN ≤ ULN
   * AST ≤ ULN
   * ALT ≤ ULN
   * Alkaline Phosphatase ≤ ULN
   * Total Bilirubin < 1.5 x ULN AND Direct Bilirubin ≤ ULN
   * HgbA1c ≤ 6.4

Exclusion Criteria:

1. Previous receipt of humanized or human monoclonal antibody whether licensed or investigational.
2. Positive serology for HIV antibody, HCV antibody or Hepatitis B surface antigen.
3. Regular use of more than 20 cigarettes per day (or equivalent amount of nicotine containing product)
4. Drug or alcohol abuse within previous 12 months or a positive screen within 24 hours of study product administration.
5. History of a previous severe allergic reaction with generalized urticaria, angioedema or anaphylaxis.
6. Any current medical or other condition that in the opinion of the PI would jeopardize the safety of the volunteer participating in the study.
7. Clinically significant gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, or infectious disease, as determined by the PI. The investigator will consider all conditions, which could conceivably increase risk to the subjects, alter study drug metabolism, or jeopardize data integrity as clinically significant when making this determination.
8. Physical finding on examination considered clinically significant such as murmur (other than functional), hepatosplenomegaly, lymphadenopathy or focal neurological deficit.
9. Positive serum pregnancy test during screening or within 24 hours of study product administration, or an unwillingness to undergo pregnancy testing.
10. Breast-feeding.
11. Treatment with another investigational drug or other investigational intervention within 30 days of study drug dosing.
12. Safety laboratory abnormalities at Screening or Day -1, which are clinically significant as determined by the PI.
13. Tick bite within 4 weeks prior to screening.
14. Receipt of any Lyme disease vaccine.

Abnormal ECG or laboratory parameters may be repeated once, if in the opinion of the PI, the results are due to technical factors or are inconsistent with the potential subject's medical evaluation.

Potential study subjects who met all inclusion and none of the exclusion criteria, but who, for personal or administrative reasons, were not included in a study cohort, may be rescreened if more than 30 days have passed since their previous screening. There are no restrictions on the number of re-screens permitted for these subjects.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a study treatment by number of adverse events reported | Day 1 through Day 360
  Adverse events will be assessed by targeted medical history, physical examination, and laboratory testing. Abnormal laboratory values constitute adverse events only if they induce signs or symptoms and/or require therapy that are new or enhanced from baseline. Injection site reactions (pain, tenderness, erythema/redness, and induration/swelling) will be evaluated pre-dose through Day 15. The reactions are rated Mild (Grade 1), Moderate (Grade 2), and Severe (Grade 3) according to FDA guidance for industry. Adverse events will be summarized by System Organ Class (SOC) using MedDRA.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter: Maximum serum concentration observed (Cmax) of 2217LS | 14 Study Days - Day-1 Pre Dose, Day 2 or 3, 4 or 5, 6 or 7, 8 or 9, 10 or 11, 14 or 15, 29, 60, 90, 120, 180, 240, 360
  Serial measurements of 2217LS concentration in the serum.
Pharmacokinetics (PK) parameter: Area under the curve (AUC) of 2217LS | 14 Study Days - Day-1 Pre Dose, Day 2 or 3, 4 or 5, 6 or 7, 8 or 9, 10 or 11, 14 or 15, 29, 60, 90, 120, 180, 240, 360
  Serial measurements of 2217LS concentration in the serum.
Pharmacokinetics (PK) parameter: Serum half life (T 1/2) of 2217LS | 14 Study Days - Day-1 Pre Dose, Day 2 or 3, 4 or 5, 6 or 7, 8 or 9, 10 or 11, 14 or 15, 29, 60, 90, 120, 180, 240, 360
  Serial measurements of 2217LS concentration in the serum.
Assessment of immunogenicity anti-drug antibodies (ADA) of 2217LS | 10 Study Days - Day 1 Pre-Dose, Day 8 or 9, 14 or 15, 29, 60, 90, 120, 180, 240, 360
  Serial measurements of 2217LS concentration in the serum.

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion Inc., Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No